CLINICAL TRIAL: NCT02171182
Title: A Non-interventional Post-registration Clinical Study of Efficacy and Safety of Qutenza in Patients With Post-operative Peripheral Neuropathic Pain
Brief Title: A Study of Efficacy and Safety of Qutenza in Patients With Post-operative Peripheral Neuropathic Pain
Status: Completed | Type: Observational
Sponsor: Astellas Pharma s.r.o. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 0805-MA-1001
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Post-operative Peripheral Neuropathic Pain
Keywords: Qutenza; 8% capsaicin patch; Non-interventional; Post-operative peripheral neuropathic pain; Observational; Czech Republic
MeSH Terms: interventions — Capsaicin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Qutenza patients w/ post-operative peripheral neuropathic pain
  Interventions: Drug: Qutenza

INTERVENTIONS:
Drug: Qutenza — capsaicin patch
  Other Names: NGX-4010,; A0805,; Capsaicin

SUMMARY:
The aim of this study is to monitor the effectiveness and used dosage of the 8% capsaicin patch in real-life clinical practice in the treatment of post-operative neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed peripheral post-operative neuropathic pain

Exclusion Criteria:

* hypersensitivity to capsaicin
* pregnancy
* diabetes mellitus
* treatment of face

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with post-operative peripheral neuropathic pain
Sampling Method: Probability Sample
Enrollment: 319 (Actual)
Dates: Start 2014-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Percentage rate of responders | Baseline, Week 13
  at least 30% decrease in pain intensity as compared to the baseline

SECONDARY OUTCOMES:
Basic demographic parameters | Baseline
  age, gender, history of the disease, other diagnoses
Previous treatment of neuropathy | Baseline
  type of treatment, dosage, combination, treatment line number
Reason for a change in the therapy | Baseline
Dose | Baseline, Week 13 and Week 26
  number of patches, area of application and frequency of treatment with 8% capsaicin
Size of the area affected by neuropathic pain | Baseline, Week 13 and Week 26
Concomitant neuropathic medication | Baseline, Week 13 and Week 26
Efficacy of treatment | Baseline, Week 8, Week 13 and Week 26
  changes in NPRS score between weeks 0 and week 8, week 13 and week 26
Quality of life questionnaire (EQ-5D) | Baseline, Week 8, Week 13 and Week 26
Consumption of rescue analgesic medication | Baseline, Week 8, Week 13 and Week 26
Consumption of additional medical care for neuropathic pain | Baseline, Week 8, Week 13 and Week 26
  extra visits, hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Medical and Scientific Affairs manager, Study Director — Astellas Pharma s.r.o.
Locations (29):
- Czechia (29):
  - Site CZ42019 Hospital, Benešov
  - Site CZ42026 Hospital, Beroun
  - Site CZ42008 Onco Clinic, Brno
  - Site CZ42001 Sv. Anna Hospital, Brno
  - Site CZ42007 Private Practice, České Budějovice
  - Site CZ42015 Hospital, Havlíčkův Brod
  - Site CZ42029 Hospital, Hořovice
  - Site CZ42009 University Hospital, Hradec Králové
  - Site CZ42004 Hospital, Jihlava
  - Site CZ42022 Hospital, Karlovy Vary
  - Site CZ42017 Hospital, Klatovy
  - Site CZ42025 Private Practice, Krnov
  - Site CZ42016 Hospital, Liberec
  - Site CZ42023 Hospital, Mladá Boleslav
  - Site CZ42020 Hospital, New Town
  - Site CZ42010 University Hospital, Olomouc
  - Site CZ42012 Hospital, Opava
  - Site CZ42002 University Hospital, Ostrava
  - Site CZ42006 University Hospital, Pilsen
  - Site CZ42013 Hospital, Prague
  - Site CZ42018 Rheumatological Institute, Prague
  - Site CZ42005 University Hospital, Prague
  - Site CZ42021 Military Hospital, Prague
  - Site CZ42027 Hospital, Semily
  - Site CZ42011 Hospital, Sokolov
  - Site CZ42024 Hospital, Teplice
  - Site CZ42028 Hospital, Uherské Hradiště
  - Site CZ42014 Private Practice, Vysoké Mýto
  - Site CZ42003 Bata Hospital, Zlín

IPD SHARING:
Plan to Share IPD: Undecided